CLINICAL TRIAL: NCT04833179
Title: Fecal Transplant for Alopecia Areata
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Eli Sprecher, MD, Liat Samuelov MD. Vice Chair, Division of Dermatology, Tel Aviv Sourasky Medical Center, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 001320
Record Dates: First submitted 2021-03-01; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Fecal transplant; Microbiome
MeSH Terms: conditions — Alopecia Areata | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: 110 patients with alopecia areata.
  Prior the beginning of the study all subjects will undergo:
  Complete physical examination Clinical image of involved locations will be taken Estimating the severity of the disease Microbiome samples Blood sample
  The patients with AA will undergo randomization into two groups. Group 1 - the subjects will receive a complete fecal transplant course. Group 2 - the subjects will receive placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fecal transplant (Experimental): Healthy donors will be selected by the fecal transplant unit, in Tel-Aviv medical center. The treatment will be given in the form of fecal capsule. Each capsule will contain a double capsule with 2 layers to ensure that the fecal material will be contained. The treatments will include 30 capsules for the first treatment, that will be taken in two consecutive days, each day 15 capsules. The second, third and fourth treatments will all include 15 fecal capsules. There will be 2 weeks intervals between each treatment.
  Interventions: Biological: fecal transplant
- placebo (Placebo Comparator): Placebo capsule that can not be differentiate from the focal transplant capsule will be given in the same interval as the fecal transplant procedure written above.
  Interventions: Other: placebo

INTERVENTIONS:
Biological: fecal transplant — Healthy donors will be selected by the fecal transplant unit, in Tel-Aviv medical center. All donors will undergo a screening process that will include a detailed medical history, blood work and fecal tests. Only after passing the screening, the donor will be added to the groups of donors that will participant in this study.
  The treatment will be givenin the form of fecal capsule. Each capsule will contain a double capsule with 2 layers to ensure that the fecal material will be contained. The treatments will include 30 capsules for the first treatment, that will be taken in two consecutive days, each day 15 capsules. The second, third and fourth treatments will all include 15 fecal capsules. There will be 2 weeks intervals between each treatment.
  Arms: fecal transplant
Other: placebo — placebo
  Arms: placebo

SUMMARY:
the investigators intend to analyze the microbiome in the diseased areas, healthy skin and fecal samples. In addition, the investigators plan to evaluate how the fecal transplant can influence the severity of the disease and hair growth, all in hope that fecal transplant can help to treat or even cure AA. This may help dermatologists in the future and expand the treatment options for AA.

DETAILED DESCRIPTION:
Alopecia areata (AA) is a common autoimmune disease that triggers non scarring hair loss in different severities. Usually the hair loss will be contained to the scalp and / or beard, but in some cases, there will be total hair loss from the entire scalp (alopecia totalis), or complete loss of all body, facial and scalp hair (alopecia universalis).

AA is an autoimmune disease that produces an inflammation surrounding the hair follicles, this leads to temporary hair loss. In cases the disease become chronic, the immune system attack may lead to a permanent hair loss. This common hair disease has a significant impact on the patient's quality of life, it can cause impairment on the patient's confidence, self-esteem, lead to depression and more.

Lately two patients with AA and clostridium difficile infection were treated with fecal transplantation for their infection (Rebello et al. 2017). After the transplant a significant improvement was notice in hair growth. These 2 cases raised the option that a fecal transplant may have an additional effect on the autoimmune reaction against the hair follicle in AA.

the investigators intend to analyze the microbiome in the diseased areas, healthy skin and fecal samples. In addition, the investigators plan to evaluate how the fecal transplant can influence the severity of the disease and hair growth, all in hope that fecal transplant can help to treat or even cure AA. This may help dermatologists in the future and expand the treatment options for AA.

ELIGIBILITY:
Inclusion Criteria:

AA patients with:

* Acute disease that appeared in the last 3 months.
* Recurrence of AA in the last 3 months, in a patient who had remission for at least one year.
* At least one patch of hair loss on the scalp and / or the beard, or with a widespread disease such as total loss of the hair over the entire scalp (alopecia totalis).
* In case of a single alopetic patch, the patch must be equal or bigger than 2 cm in diameter.
* All patients will be diagnosed by two separate dermatologist, or one dermatologist with the support of classical finding on skin biopsy.

Exclusion Criteria:

1. Patients who were treated with systemic corticosteroids / corticosteroids injection one year prior the study.
2. Patients who were treated with topical corticosteroids two weeks prior the study.
3. Patients who were treated with immunosuppressing medications or biological treatments one year prior the study.
4. Patients who were treated with systemic antibiotics of any kind 3 months prior the study.
5. Patient who were treated with topical antibiotics one months prior the study.
6. Patients who were treated with probiotics one months prior the study.
7. Patients with alopecia universalis (total loss of all body, scalp and facial hair).
8. Patients with bowel disease or an active infection including clostridium difficile.
9. Pregnant and breastfeeding women.
10. Childrenbelow the age of 18.
11. Malignant disease in the past 5 years.
12. Patient with any infectious disease that require antibiotics during the study period.

In any case a patient would like to withdraw from the study, for any reason, all samples will be destroyed immediately, and the patient will stop his participant in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Severity alopecia tool score - SALT score I | up to1 year after fecal transplantation
  The SALT score I (Olsen, 2004) is a global severity score that captures percentage hair loss.
  The scalp area is divided into 4 quadrants - Left (L) Right (R) Back (B) Top (T). Photographs taken of the four views of the scalp. The percentage of hair loss in any one of the four views (areas) of the scalp = the percentage hair loss X percent surface area of the scalp in that area.
  1. left side view = ALOPECIA% x 18%
  2. right side view = ALOPECIA% x 18%
  3. top of scalp = ALOPECIA% x 40%
  4. back of scalp = ALOPECIA% x 24% The SUM of all equals the score. (possible score range: 0-100)
Alopecia Areata Progression Index, AAPI | up to1 year after fecal transplantation
  formula for the total AAPI score (possible score range: 0-600). The scalp area is divided into 4 quadrants - Left (L) Right (R) Back (B) Top (T) using the Olsen/Canfield tool. The percent alopecic area (%AA) and score of hair loss activity (SL) is determined in each quadrant.
  The %AA is defined as the percentage of alopecic area in each compartment. SL is calculated as the sum of the results of hair pull tests (2 = positive, excessive, i.e. >20% of grasped hairs; 1 = positive, not excessive, 10-20%; 0 = negative, <10%) and the magnification findings associated with hair loss activity such as exclamation mark hairs, broken hairs and black dots (4 = ≥50%, 2 = <50%, 0 = 0%) in each quadrant.
  The total AAPI score is calculated by the following formula:
  [%AA(L) × SL(L) × 0.18] + [%AA(R) × SL(R) × 0.18] + [%AA(T) × SL(T) × 0.4] + [%AA(B) × SL(B) × 0.24].
  (possible score range: 0-600)
patient assessment. | up to1 year after fecal transplantation
  1. <25% regrowth.
  2. 25%<x<50% regrowth.
  3. 50%<x<70%regrowth.
  4. >75% regrowth.
  5. 100% regrowth.

CONTACTS AND LOCATIONS:
Overall Officials: Liat Samueluv, MD, Principal Investigator — Vice chair, Department of Dermatology Tel Aviv Sourasky Medical center, Israel

IPD SHARING:
Plan to Share IPD: No